CLINICAL TRIAL: NCT01317927
Title: A Phase I Study of Belinostat in Combination With Warfarin in Patients With Solid Tumors or Hematological Malignancies
Brief Title: A Study of Belinostat in Combination With Warfarin in Patients With Solid Tumors or Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-CLN-20
Record Dates: First submitted 2011-03-09; First posted 2011-03-17 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Solid Tumor; Hematological Malignancy
Keywords: belionstat; warfarin; hematological malignancy; solid tumors; PK/PD study
MeSH Terms: conditions — Hematologic Neoplasms | interventions — belinostat; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Warfarin, Belinostat (Experimental): Warfarin 5 mg po will be given on Day -14 and Day 3. Belinostat 1000 mg/m² will be given as a 30 minute IV infusion on Days 1 - 5
  Interventions: Drug: Belinostat, Warfarin

INTERVENTIONS:
Drug: Belinostat, Warfarin — 1000 mg/m2 injection infusion given in a 30 min period plus Warfarin 5mg PO
  Other Names: PXD101

SUMMARY:
The purpose of this study is to evaluate the plasma concentration and pharmacodynamics effects of warfarin 5 mg, in the presence or absence of belinostat 1,000 mg/m².

Pharmacokinetic evaluation of belinostat 1,000 mg/m² and metabolites in the presence of warfarin 5 mg.

DETAILED DESCRIPTION:
This is an open-label, single center, pharmacokinetic and pharmacodynamic study in patients with solid tumor or hematological malignancies. Upon providing informed consent and satisfying screening procedures, eligible subjects will report to the clinic for Part I of the study 14 days before the first dose of belinostat (Day -14) for clinical laboratory tests, warfarin (5mg) single dose and a series PK collections. On days 1-5 of each 21-day cycle patients will receive belinostat 1000mg/m*2 and will have a series of subsequent PK samples collected. On day 3 of cycle 1 only, the patient will also receive warfarin 5mg single dose prior to belinostat infusion. PK samples, urine samples, electrocardiogram (ECG) and safety measurements will be collected from Day 1 through Day 10 of cycle one. If it is in the interest of the patient, belinostat can be continued during Part II- extension phase for 5 additional cycles of belinostat treatment on days 1-5 of each subsequent cycle, or until disease progression, patient withdraws consent or if unacceptable toxicity occurs. During the extension phase routine physical exams, laboratory tests and safety and efficacy assessments will be performed. Disease evaluations will be conducted per standard of care. Patients who discontinue for reasons other than disease progression will be followed until new anti-cancer treatment is initiated or death.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histological or cytological confirmed diagnosis of malignant disease
* Age ≥18 years old
* Adequate organ function
* ECOG 0-2
* Estimated life expectancy >3months
* Negative pregnancy test for women of child bearing potential

Exclusion Criteria:

* Low dose anticoagulation therapy within 2 week prior to study treatment
* Anticancer therapy within 2 weeks prior to study treatment
* Investigational therapy within 4 weeks of study treatment
* Major surgery within 2 weeks of study treatment
* Coexisting active infection or other medical condition likely to interfere with trial procedures
* Significant cardiovascular disease (NYHA Class III or IV)
* Baseline prolongation of QT/QTc
* Clinically significant CNS disorder, altered mental status or psychiatric disorders precluding understanding of the informed consent process and/or completing trial procedures
* Symptomatic or untreated CNS metastases
* Pregnant or breast feeding women
* Patients not willing to use effective contraception
* Known infection with HIV, Hep B or Hep C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentration and pharmacodynamic effects of warfarin | 34 days
  Samples will be analyzed for S-warfarin and R-warfarin analytes in all evaluable subjects at the end of the trial
Pharmacokinetic evaluation of belinostat | 34 days
  Pharmacokinetic evaluation of belinostat 1,000 mg/m2 and metabolites in the presence of warfarin 5mg

SECONDARY OUTCOMES:
Presence of PK analytes for all subjects. | 34 days
  To measure the following analytes of all evaluable subjects at the end of the trial: Belinostat, belinostat glucuronide, methylated belinostat, Beliostat amide, belinostat acid and 3-ASBA.
Safety profile of belinostat given concomitantly with warfarin | 34 days
  To evaluate the safety profile of belinostat given concomitantly with warfarin 5mg. Safety and tolerability assessment include adverse events (AEs), physical examination, vital signs, clinical laboratory tests, and electrocardiograms (ECGs).
Overall survival of patients | 8 months
  To evaluate progress-free survival and to assess tumor measurement

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, FACP, Principal Investigator — Huntsman Cancer Institute, University of Utah, 2000 Circle of Hope, UT 84112
Locations (1):
- Huntsman Cancer Center, University of Utah, Salt Lake City, Utah, United States